CLINICAL TRIAL: NCT07251374
Title: Construction of a Multicenter Disease-Specific Database and Prospective Cohort for Osteomyelitis
Brief Title: Osteomyelitis Multi-center Prospective Cohort Study
Status: Not yet recruiting | Type: Observational
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Dong Sun, Associate Professor, Southwest Hospital, China
Other Study IDs: (A)KY2025236
Record Dates: First submitted 2025-11-17; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Osteomyelitis of Lower Extremities
Keywords: Osteomyelitis; Multi-center; Prospective; Disease-Specific Database
MeSH Terms: conditions — Osteomyelitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgically Treated Cohort: All treatments will be conducted in accordance with existing clinical practice guidelines. This study is purely observational; it will only monitor and collect data on changes in relevant parameters during the subjects' treatment process without interfering with any other clinical decisions.
  Enrolled subjects will be assigned to different treatment regimens based on their diagnosis and differential diagnosis. Patients with bone infection who do meet the criteria for surgical intervention will receive conservative therapy.
- Conservatively Treated Cohort: All treatments will follow current standards of care. This is an observational study that collects data on treatment outcomes without intervening in clinical management. Patients who meeting the surgical indications will undergo surgical treatment.

SUMMARY:
To establish a prospective, multicenter, real-world cohort of patients with osteomyelitis, by systematically collecting and analyzing detailed treatment and follow-up data, in order to provide clinical evidence for the standardization of its treatment

DETAILED DESCRIPTION:
Study Design： This is a prospective, multi-center, real-world clinical study. Subjects will be assigned to different treatment regimens based on their diagnosis and differential diagnosis.

Conservatively Treated Cohort: Patients with bone infection who do not meet the criteria for surgical intervention will receive conservative therapy, which includes intravenous (IV) and oral antibiotics.

Surgically Treated Cohort: Patients meeting the surgical indications will undergo a staged surgical protocol. The first stage involves debridement and implantation of antibiotic-impregnated bone cement. The need for auxiliary internal or external fixation will be determined based on the patient's condition. The second stage, performed 8 weeks after the first, focuses on repairing the bone defect.

All treatments will be conducted in accordance with current clinical practice guidelines. This study is purely observational; it will only monitor and collect data on changes in relevant parameters during the treatment process without interfering with any other clinical decisions.

Data Collection：

The following information will be recorded and collected:

1. Unique subject identifier and basic demographic information.
2. Baseline status and information prior to treatment.
3. Key information related to the surgery.
4. Post-operative follow-up information, including:

（1）Pain score (Visual Analog Scale, VAS) （2)Quality of life (Short Form-36, SF-36) (3)Self-Rating Anxiety Scale (SAS) score (4)Limb function score (Disabilities of the Arm, Shoulder and Hand / Lower Extremity Functional Scale, DASH/LEFS) (5)Range of motion of adjacent joints (6)Occurrence of complications.

Complications include:

1. Surgical incision complications (e.g., dehiscence, skin necrosis).
2. Pin tract infection.
3. Fixation failure or breakage.
4. Reduced joint range of motion.
5. Other discomforts deemed by the investigator to be related to the surgery.

Cohort Stratification:

To comprehensively describe the clinical characteristics and outcomes of bone infection, the study data will be stratified into cohorts based on the real-world treatment received by the patients. Patients will be categorized into cohorts according to the actual treatment modality they received, with each treatment type constituting a separate cohort. All cohort classifications will be performed after data collection is complete, based on predefined criteria, and will not involve proactive intervention by the investigators.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent provided.
2. Diagnosis of osteomyelitis confirmed by the site per guidelines (including definitive/suggestive criteria).

Exclusion Criteria:

1. Patients who, in the opinion of the investigator, are unable to comply with the entire study procedure (including postoperative management and regular follow-up) due to psychiatric, cognitive, or behavioral disorders, or other objective reasons.
2. Any other condition that, in the opinion of the investigator, would make the patient unsuitable for participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of real-world patients with osteomyelitis from multiple centers. Based on the treatment received, participants will be retrospectively assigned to either a conservative therapy cohort or a surgical therapy cohort for analysis.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Infection control rate at week 8 after treat | 8 weeks after operation
  Patients will return for a follow-up visit at 8 weeks post-treatment. The assessment will include evaluation of the incision condition, documentation of afebrile status, and repeat laboratory tests including CBC (WBC count), ESR, and CRP

SECONDARY OUTCOMES:
Disability of Arm Shoulder and Hand Scale（DASH） | Pre-treatment; At 8 weeks post-treatment; At 12 months post-treatment
  This outcome measure is applicable only to patients presenting with upper extremity symptoms or dysfunction.Patients will be guided by study staff to complete the questionnaire based on their actual condition.
  Disability of Arm Shoulder and Hand Scale（DASH）：
  1. Scoring: The total score ranges from 0 to 100.
  2. Interpretation: A score of 0 indicates no disability (normal upper extremity function), while a score of 100 indicates severe disability (extremely limited upper extremity function).
The 36-Item Short Form Health Survey | Pre-treatment; At 8 weeks post-treatment; At 12 months post-treatment
  Patients will be guided by study staff to complete the questionnaire based on their actual condition.
  1. Scoring: The total score ranges from 0 to 900.
  2. Interpretation:The 36-Item Short Form Health Survey（SF-36）assesses health status across nine dimensions: Physical Functioning (PF), Role-Physical (RP), Bodily Pain (BP), General Health (GH), Vitality (VT), Social Functioning (SF), Role-Emotional (RE), Mental Health (MH), and Health Transition (HT). For all scales, higher scores indicate a better health status for the respondent.
Self-Rating Anxiety Scale (SAS) | Pre-treatment; At 8 weeks post-treatment; At 12 months post-treatment
  Patients will be guided by study staff to complete the questionnaire based on their actual condition.
  1. Scoring: The total score ranges from 0 to 80.The standard cutoff for anxiety is a score of 50.
  2. Interpretation:Mild anxiety: 50-59；Moderate anxiety: 60-69；Severe anxiety: 70 and above.
Pain score (assessed by Visual Analogue Scale) | Pre-treatment;At 2 weeks post-treatment; At 8 weeks post-treatment; At 12 months post-treatment
  Patients will be guided by study staff to complete the questionnaire based on their actual condition.
  1. Scoring: The total score ranges from 0 to 10.
  2. Interpretation: A score of 0 indicates "No Pain"；A score of 10 indicates "The Worst Possible Pain" (or "Severe/Excruciating Pain").
Lower Extremity Functional Scale | Pre-treatment; At 8 weeks post-treatment; At 12 months post-treatment
  This outcome measure is applicable only to patients presenting with lower extremity symptoms or dysfunction. Patients will be guided by study staff to complete the questionnaire based on their actual condition.
  Lower Extremity Functional Scale（LEFS）：
  1. Scoring: The total score ranges from 0 to 80.
  2. Interpretation: A higher score indicates a higher level of lower extremity function. Conversely, a lower score indicates greater functional limitation.

CONTACTS AND LOCATIONS:
Overall Officials: Dong Sun, MD, Principal Investigator — The First Hospital Affiliated of Army Medical University
Locations (1):
- The First Hospital Affiliated to Army Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: January 2030-January 2031
Access Criteria: Data will be shared with qualified researchers who submit a methodologically sound proposal. Proposals must be directed to sumersun07@126.com. A data access agreement (DAA) must be signed. Data will be de-identified and the requestor must agree to the terms and conditions of the DAA, which include commitments to: 1) using the data only for the specified research purpose, 2) securing the data using appropriate computer technology, 3) destroying the data after analysis, and 4) not attempting to identify any individual participant. Requests for data will be reviewed by an internal review committee to ensure scientific validity and that the use of data is consistent with the informed consent provided by study participants.